CLINICAL TRIAL: NCT05446428
Title: Evaluation of Type I IFN Level and Disease Activity in SLE Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: V.A. Nasonova Research Institute of Rheumatology, Moscow (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Popkova Tatiana, MD PhD Professor, V.A. Nasonova Research Institute of Rheumatology, Moscow
Other Study IDs: D3461L00006
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Elevated Level of IFN Type I in SLE Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Any SLE Disease Activity
  Interventions: Other: study of IFNGS expression biomarkers
- Moderate to severe SLE Disease Activity
  Interventions: Other: study of IFNGS expression biomarkers

INTERVENTIONS:
Other: study of IFNGS expression biomarkers — Blood tests for serum biomarkers, autoantibodies, cytokine profile etc.

SUMMARY:
Elevated level of IFN type I in SLE patients associated with certain serum biomarkers (galectin -1,-3,-9; cytokine profile - 20 plex panel - GM-CSF, IFN-γ, IL-2, -4,-5,-6,-7,-8,-10,-13,-15,-17,-18, IP-10. MCP-1, MIG, MIP-1α, MIP-1β, RANTES, TNF-α, TNF-RII, BAFF, APRIL), clinical and laboratory manifestations, activity and duration pf the disease and SLE patients quality of life. Standard immunosuppressive and anti-B-cell therapy can reduce the IFN type I and associated biomarkers levels in patients with high and moderate disease activity (SLEDAI-2К ≥6).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years old
2. Patients with SLE (SLICC/ACR 2012) confirmed by rheumatologist
3. Provided written informed consent before any study-related procedures are performed.
4. Ability to attend scheduled visits
5. No positive changes in the course of standard of care SLE therapy (glucocorticoids in stable doses, hydroxychloroquine and/or immunosuppressant therapy) at least 30 days before screening.

Exclusion Criteria:

1. Participation in any other clinical study
2. Pregnancy or pregnancy planning in next 12 months, lactation
3. Acute infectious disease or relapse of chronic infectious disease.
4. Receiving any of biologic agent or Janus-kinases inhibitors during 24 months prior to screening.
5. Active severe or unstable neuropsychiatric SLE manifestations (convulsion, psychosis, delirium, hallucinations, coma, transverse myelitis).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 70 adult patients with SLE who receive inpatient or outpatient саre from 01.06.2022 (1 stage) 30 of them with moderate to severe disease activity (SLEDAI 2К ≥6) will be included in prospective observation (2 stage 01.06.2022-25.12.2023)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Pathogenetic, clinical and prognostic significance of IFN stimulated genes expression - IFNGS biomarkers in SLE patients | Sept 1 2022 - Nov 1 2022
  Pathogenetic, clinical and prognostic significance of IFN stimulated genes expression - IFNGS biomarkers (IFI44L, MX1, IFIT 1, RSAD2, EPSTI1), serum biomarkers (galectin -1,-3,-9; cytokine profile - 20 plex panel - GM-CSF, IFN-γ, IL-2, -4,-5,-6,-7,-8,-10,-13,-15,-17,-18, IP-10. MCP-1, MIG, MIP-1α, MIP-1β, RANTES, TNF-α), TNF-α receptors type II (TNF-RII), В-cell activation factors (BAFF, APRIL) in SLE patients.

SECONDARY OUTCOMES:
Rate of IFN stimulated genes | Nov 1 2022 - Oct 31 2024
  Rate of IFN stimulated genes hyper-expression, serum biomarkers level (galectin -1,-3,-9; cytokine profile - 20 plex panel - GM-CSF, IFN-γ, IL-2, -4,-5,-6,-7,-8,-10,-13,-15,-17,-18, IP-10. MCP-1, MIG, MIP-1α, MIP-1β, RANTES, TNF-α), TNF-α receptors type II level (TNF-RII), В-cell activation factors level (BAFF, APRIL) in SLE patient's blood.
IFN stimulated genes hyper-expression and serum biomarkers level | Nov 1 2022 - Oct 31 2024
  IFN stimulated genes hyper-expression and serum biomarkers level (galectin -1,-3,-9; cytokine profile - 20 plex panel - GM-CSF, IFN-γ, IL-2, -4,-5,-6,-7,-8,-10,-13,-15,-17,-18, IP-10. MCP-1, MIG, MIP-1α, MIP-1β, RANTES, TNF-α), TNF-α receptors type II level (TNF-RII), В-cell activation factors level (BAFF, APRIL) associated with SLE clinical and laboratory manifestations (such as muco-cutaneous, joints, renal, hematological, immunological et ctr.), disease activity (assessed with SLEDAI-2k) and duration, patients' quality of life.
IFNGS | Nov 1 2022 - Oct 31 2024
  IFNGS alone or as a part of complex poly-parametric indexes is a predictor of standard immunosuppressive and anti-B-cell therapy effectiveness in SLE and flares prevention.

IPD SHARING:
Plan to Share IPD: No